CLINICAL TRIAL: NCT01056211
Title: 1540nm Non Ablative Fractional Laser Treatment of Scars : a Prospective Single Blinded Within Patient Controlled Randomized Trial.
Brief Title: 1540nm Non Ablative Fractional Laser Treatment of Scars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/626
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix | interventions — Laser Therapy; Therapeutics; Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- hypopigmented scars treated with laser (Active Comparator): patients with hypopigmented scars treated with Starlux 300 Lux 1540nm Fractional laser hand piece
  Interventions: Procedure: laser treatment
- hypopigmented scars treated without laser (Placebo Comparator): patients with hypopigmented scars treated without laser
  Interventions: Procedure: treatment without laser
- hypertrophic scars treated with laser (Active Comparator)
  Interventions: Procedure: laser treatment
- hypertrophic scars not treated with laser (Placebo Comparator)
  Interventions: Procedure: treatment without laser
- scars due to grafts and reconstructions treated with laser (Active Comparator): scars due to grafts and reconstructions in the head and neck region
  Interventions: Procedure: laser treatment
- grafts and reconstructions scars not treated with laser (Placebo Comparator): scars due to grafts and reconstructions in the head and neck region
  Interventions: Procedure: treatment without laser

INTERVENTIONS:
Procedure: laser treatment — Starlux 300 Lux 1540nm Fractional laser hand piece
  Arms: hypertrophic scars treated with laser; hypopigmented scars treated with laser; scars due to grafts and reconstructions treated with laser
Procedure: treatment without laser — Starlux 300 Lux 1540nm Fractional laser hand piece
  Arms: grafts and reconstructions scars not treated with laser; hypertrophic scars not treated with laser; hypopigmented scars treated without laser
Procedure: laser treatment — Starlux 300 Lux 1540nm Fractional laser hand piece
  Arms: scars due to grafts and reconstructions treated with laser

SUMMARY:
Scars are a frequent reason of consultation in a dermatological clinic. Their cosmetic aspect can play a key role in patient satisfaction and self-image.

Non ablative fractional infra-red laser treatment is a new concept in the laser field using arrays of microscopic thermal damage patterns to stimulate a wound healing response. There are different reports on the positive effect of these type of laser treatment in the treatment of acne scarring, striae, rythides, hypopigmented and hypertrophic scars.

The low morbidity of the treatment and the lack of satisfying treatment regimes for different types of scars makes it attractive to investigate the efficacy and safety of 4 treatment with the 1540nm non ablative fractional laser in the treatment of scars.

Objectives:

* To evaluate the efficacy of 4 laser treatments with Starlux 300 Lux 1540nm Fractional laser handpiece ( Palomar Medical Technologies ) 1 and 3 month after the last laser treatment for 3 different "scar" patient groups :

  1. Patients with hypopigmented scars
  2. Patients with hypertrophic scars
  3. Patients with scars due to grafts and reconstructions in the head and neck region.
* To evaluate the treatment related pain. on a categorical scale from 0-10
* To evaluate the adverse effect of 1540nm fractional laser versus untreated control in the 3 patient groups.

The study design is a prospective single blinded randomised within-patient controlled study The study involves 6 visits.

ELIGIBILITY:
The patients needs to have a scar fulfilling the inclusion and exclusion criteria of one of the 3 patient groups:

Patient group 1: patients with hypopigmented scars :

Inclusion criteria:

* Patients with a hypopigmented scar allowing 2 side by side test areas of similar sizes and appearance within the same anatomical region.
* Skin type 1-4
* Age at least 18 years old
* Willingness and ability to give written informed consent and to comply with the requirements of the protocol

Exclusion criteria:

* Pregnancy and lactation
* Oral retinoid drugs within the past 6 months

Patientgroup 2: patients with hypertrophic scars :

Inclusion criteria:

* Patients with a hypertrophic scar allowing 2 side by site test areas of similar sizes and appearance within the same anatomical region.
* Skin type 1-4
* Male / Female
* Age at least 18 years old
* Willingness and ability to give written informed consent and to comply with the requirements of the protocol

Exclusion criteria:

* Pregnancy and lactation
* Oral retinoid drugs within the past 6 months

Patient group 3: Patients with scars due to grafts and reconstructions in the head and neck region.

Inclusion criteria:

* Patients with a graft or reconstruction with 2 site by site test areas of similar sizes and appearance within the same anatomical region (head and neck region).
* Skin type 1-4
* Age at least 18 years old
* Willingness and ability to give written informed consent and to comply with the requirements of the protocol

Exclusion criteria:

* Pregnancy and lactation
* Oral retinoid drugs within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
efficacy of 4 laser treatments with Starlux 300 Lux 1540nm Fractional handpiece (Palomar Medical Technologies) 1 and 3 months after the last laser treatment in 3 different "scar" patient groups | at 1 and 3 months
Evaluation of the treatment related pain | at 1 and 3 months
Evaluation of the adverse effect of 1540nm fractional laser versus untreated control site | at 1 and 3 months

SECONDARY OUTCOMES:
Evaluation of skin redness and pigmentation | at 1 and 3 months after treatment
Compare different clinical scar assessment tools that can be used in the evaluation of clinical efficacy of the laser treatment | at 1 and 3 months after treatment
Physician assessment for the treated and control region (PhGA) | at 1 and 3 months after treatment
patient assessment for the treated and control region | at 1 and 3 months after treatment
Photografic documentation of scar improvement | at 1 and 3 months after treatment
Evaluation of histological difference in treated an non treated parts of the scar | at 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Verhaeghe, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Univerisity Hospital Ghent, Ghent, Belgium